CLINICAL TRIAL: NCT05922293
Title: Combined Effects of Blow Bottle Technique and Percussion Technique in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Combined Effects of Blow Bottle Technique and Percussion Technique in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0320
Record Dates: First submitted 2023-06-06; First posted 2023-06-28 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Airway Obstruction; COPD; Dyspnea; Expiratory flow rate; Percussion.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Airway Obstruction; Dyspnea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blow Bottle technique (Active Comparator): Blowing with a straw into a water bottle is a good exercise to improve breathing capacity. The user, who has poor pulmonary function, always has his "blow bottle" handy
  Interventions: Other: blow bottle
- percussion (Experimental): Percussion technique should be performed for about 30 seconds and simultaneously with no more than three or four lower thoracic expansion exercises
  Interventions: Other: blow bottle; Other: percussion

INTERVENTIONS:
Other: blow bottle — When you blow through a tube into water in a bottle, the pressure in the airways increases. This opens up the passageways between bronchioles, allowing air to flow behind the mucus and push it into the larger airways. This way, it will be easy to remove the mucus by coughing or huffing.
Other: percussion — Percussion technique should be performed for about 30 seconds and simultaneously with no more than three or four lower thoracic expansion exercises.
  * Do this for a total of 10 breaths,
  * Perform two huffs, and
  * Cough.
  * Close their mouth around the tube and exhale slightly forcefully for 3 seconds to produce bubbles. Such exhalations were conducted in two sets of ten, with a five-minute pause in between. For each subject, a fresh, disposable tube and bottle were utilized
  Arms: percussion

SUMMARY:
It will be a randomized control trial. Participants will be recruited according to inclusion criteria and will be allocated into 2 groups using convenience sampling technique. Group 1 will be treated with percussion technique for 30 min and group 2 with blow bottle technique combined with percussion technique for 30 min at DHQ Teaching Hospital Gujranwala. Intervention will be carried out for total 4 weeks of duration with 3 sessions per week. Outcome measures such as dyspnea, breathlessness, sputum and cough, O2 and pulse rate, expiratory flow rate will be measured by tools as mMRC, BCSS, peak flow meter respectively. Assessment will be done before and after intervention and result will be analyzed using statistical package for social sciences SPSS 20.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is characterized by nonreversible airway obstruction. A diagnosis of COPD is determined by clinical assessment of airflow limitation and symptoms such as cough and wheeze; however, the detrimental effect of COPD symptoms on a patient's quality of life (QoL) is often underestimated. Rehabilitation exercise can lessen the possibility of the progressive exacerbation of the patient's condition, exerting an active role in improving their lung function and the quality of the patients' life. Therefore, a lung function exercise bottle is designed, which is capable of adjusting the pressure according to the patient's needs. The exercise bottle is composed of three components, including bottle body, threaded round cap and air blow pipe. Furthermore, manual chest percussion is the rhythmic clapping on the chest wall with relaxed wrist and cupped hand, creating an energy wave that is transmitted to the airways. It is applied with a frequency of approximately 3-6 Hz. To reduce any adverse consequences, the technique should be performed for about 30 seconds and simultaneously with no more than three or four lower thoracic expansion exercises.

It will be a randomized control trial. Participants will be recruited according to inclusion criteria and will be allocated into 2 groups using convenience sampling technique. Group 1 will be treated with percussion technique for 30 min and group 2 with blow bottle technique combined with percussion technique for 30 min at DHQ Teaching Hospital Gujranwala. Intervention will be carried out for total 4 weeks of duration with 3 sessions per week. Outcome measures such as dyspnea, breathlessness, sputum and cough, O2 and pulse rate, expiratory flow rate will be measured by tools as mMRC, BCSS, peak flow meter respectively. Assessment will be done before and after intervention and result will be analyzed using statistical package for social sciences SPSS 20.

ELIGIBILITY:
Inclusion Criteria:

* Mild-to-Moderate COPD (according to GOLD criteria)
* Both gender (male and female)
* Aged between 35 and 80 years

Exclusion Criteria:

* Clinically unstable
* cardiovascular impairment,
* musculoskeletal dysfunction
* neurological disease

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Dyspnea (Modified Medical Research council) | fourth week
  The mMRC grade is a five-point scale based on the degree of dyspnea a patient. The use of this scale to evaluate symptoms is encouraged by current standards
Breathlessness, cough and sputum scale (BCSS) | fourth week
  In order to give a rapid and simple means of assessing the severity of respiratory symptoms frequent in COPD patients, the Breathlessness, Cough, and Sputum Scale (BCSS) was created. The BCSS is based on a three-item questionnaire that evaluates the patient's sputum production, coughing, and breathlessness
Expiratory flow rate (peak flow meter) | fourth week
  A peak flow rate should be used to capture the highest flow rates. The patient must record the highest reading out of a possible three. The best at the moment is this. A typical chart has dates with AM and PM times, a left margin, and a scale that ranges from 0 litres per minute at the bottom to 600 litres per minute at the top
O2 n pulse rate by Oximeter | fourth week
  A pulse oximeter measures the amount of oxygen that is carried by your blood. Typically, a little clip is attached to the tip of your finger. (On sometimes, the toe or earlobe are used.) A light beam is projected through the skin using the gadget. By measuring the proportion of your blood that is carrying oxygen, it calculates your oxygen level. Your oxygen saturation, often known as SpO2, is displayed on the screen

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Afzal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- DHQ Teaching Hospital, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones PW, Watz H, Wouters EF, Cazzola M. COPD: the patient perspective. Int J Chron Obstruct Pulmon Dis. 2016 Feb 19;11 Spec Iss(Spec Iss):13-20. doi: 10.2147/COPD.S85977. eCollection 2016. PMID 26937186
- [Background] Raherison C, Girodet PO. Epidemiology of COPD. Eur Respir Rev. 2009 Dec;18(114):213-21. doi: 10.1183/09059180.00003609. PMID 20956146
- [Background] Liu H, Zhang X, Zhang Y. [Design and application of a pulmonary function exercise bottle]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2019 Feb;31(2):236-237. doi: 10.3760/cma.j.issn.2095-4352.2019.02.023. Chinese. PMID 30827317
- [Background] Celli BR. Update on the management of COPD. Chest. 2008 Jun;133(6):1451-1462. doi: 10.1378/chest.07-2061. PMID 18574288